CLINICAL TRIAL: NCT02979470
Title: Study of Blood Components as Probable Prognostic and Predictive Markers of Response to Treatment in Advanced Colon and Rectal Cancers
Acronym: BMACR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: AC Camargo Cancer Center (Other)
Responsible Party: Principal Investigator, Ludmilla Thome Domingos Chinen, PhD, Principal Investigator, AC Camargo Cancer Center
Other Study IDs: CEP2141/15
Record Dates: First submitted 2016-11-29; First posted 2016-12-01 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Colon Cancer Stage IIb; Rectum Cancer, Adenocarcinoma; Colon Cancer Stage IIIa; Colon Cancer Stage IIIc; Colon Cancer Stage IIIb
Keywords: advanced colon cancer; advanced rectum cancer; circulating tumor cells; immune response; mutations
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The main reason of cancer-related mortality is the spread of cancer cells to distant sites (micrometastases). However, only a few small groups of tumor cells can metastasize by acquiring mechanism to decrease the immune response. Changes in the systemic inflammatory response to the tumor can be measured by blood-based parameters. In particular, the proportion of neutrophyls- lymphocytes (NL) has been evaluated for predicting the survival of patients with different types of cancer. The first strategy to treat colorectal cancer (CCR) is complete resection of the lesion. Nevertheless, some patients experience recurrence, probably due to residual micrometastases. We have demonstrated that analysis of some resistance proteins (Tyms / MRP1) in circulating tumor cells (CTCs) may predict treatment response in metastatic CCR patients (mCRC). We also note that the CTCs kinetics can show response to therapy. Patients with stage III disease in the colon / rectum, although showing high cure rate, generally fall locally or remotely and studies with blood markers in this group of patients is still scarce. Primary Objective: To investigate cells found in the blood (lymphocytes and neutrophils and CTCs) to verify if they can help in the choice of anti-neoplastic therapy in patients with advanced colon and rectum cancers. Secondary objectives: - to evaluate the influence of CTC kinetics in response to treatment of patients with advanced colon/rectum cancers; - to check the expression of treatment resistance, invasion and proliferation proteins (Tyms, TGF-βR, MMP-2, β-gal, Ki-67 and CD45) in CTCs and their correlation with response to treatment; - to check the mRNA expression of the same genes observed by immunocytochemistry in CTCs and their correlation with response to treatment; - to quantify CTCs, neutrophils and lymphocytes of patients included in this study and verify if there are correlation among their rates and progression-free survival. Methods: there will be collected 10 ml of blood of patients with advanced colon and rectal cancer for analysis of CTCs, lymphocytes / neutrophils. CTCs will be isolated, quantified and analyzed after separation by ISET method (Rarecells/France). The marker analysis of these cells will be done by immunocytochemistry and the gene expression will be assessed by RNAscope. The quantification of lymphocytes/neutrophils will be made by common blood count in Delboni laboratory. Expected Results: We propose to show that not only the count and the kinetics of CTCs, but also their molecular characteristics, can provide relevant information to clinicians. Hopefully, by quantification of neutrophils and lymphocytes, we will be able to identify new prognostic blood biomarkers that can direct clinicians to the best therapeutic choice.

ELIGIBILITY:
Inclusion Criteria:- ECOG (Eastern Cooperative Oncology Group) Performance Status between 0 and 2; - patients undergoing surgery followed by adjuvant chemotherapy (locally advanced colon cancer) or initiating neoadjuvant chemotherapy followed by surgery (locally advanced rectal cancer); - disease measurable by RECIST criteria 1.1 (Response Evaluation Criteria in Solid Tumors); - medullary function assessed by peripheral blood sample considered normal; Renal and hepatic function tests up to 1.5 times the limit of normality.

-

Exclusion Criteria:Patients younger than 18 years; -patients who have had surgery or surgical procedure in the last week; - patients who have had previous therapy in the last three weeks; - patients with previous history of another carcinoma in the last two years; - refuses to sign the TCLE

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: colon (EC III) or rectum (EC II and III) cancer patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 24 months
  time between first blood collection for CTC´s analysis and first progression

CONTACTS AND LOCATIONS:
Overall Officials: Ludmilla Chinen, PhD, Principal Investigator — AC Camargo Cancer Center
Locations (1):
- ACCamargo Cancer Center, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abdallah EA, Fanelli MF, Souza E Silva V, Machado Netto MC, Gasparini Junior JL, Araujo DV, Ocea LM, Buim ME, Tariki MS, Alves Vda S, Piana de Andrade V, Dettino AL, Abdon Lopes de Mello C, Chinen LT. MRP1 expression in CTCs confers resistance to irinotecan-based chemotherapy in metastatic colorectal cancer. Int J Cancer. 2016 Aug 15;139(4):890-8. doi: 10.1002/ijc.30082. Epub 2016 Apr 28. PMID 26950035
- [Result] Abdallah EA, Fanelli MF, Buim ME, Machado Netto MC, Gasparini Junior JL, Souza E Silva V, Dettino AL, Mingues NB, Romero JV, Ocea LM, Rocha BM, Alves VS, Araujo DV, Chinen LT. Thymidylate synthase expression in circulating tumor cells: a new tool to predict 5-fluorouracil resistance in metastatic colorectal cancer patients. Int J Cancer. 2015 Sep 15;137(6):1397-405. doi: 10.1002/ijc.29495. Epub 2015 Mar 11. PMID 25721610